CLINICAL TRIAL: NCT03486951
Title: Outpatient Orthognathic Surgery: "AMBOST" a One Year Prospective Study
Brief Title: Outpatient Orthognathic Surgery: "AMBOST" a One Year Study
Acronym: AMBOST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0045; 2018-A00544-51 (Other: ID-RCB)
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Orthognathic Surgery
Keywords: outpatient surgery; ambulatory surgery; length of hospital stay
MeSH Terms: interventions — Orthognathic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Orthognathic Surgery: — maxillary/mandibular osteotomies for orthognathic purposes for the treatment of a dento-maxillary dysharmony The choice between outpatient procedure or hospitalization is decided by the surgeon on a case-by-case basis according to data relating to the general state of the patient, the type of surgery, the social context, the distance from the patient's home. a medical center in accordance with the usual and legal standards of outpatient surgery

SUMMARY:
The aim of this prospective and observational study is to describe the conditions of orthognathic procedures performed in Toulouse Teaching Hospital over a one-year period, the outpatient-to-inpatient shifts rate and the whole outpatient rate among the whole orthognathic procedures done. The investigator also wants to identify factors associated with an outpatient-to-inpatient shift, and factors associated with the duration of hospitalization.

DETAILED DESCRIPTION:
In Toulouse Teaching Hospital, the annual number of orthognathic surgery outpatient stays was multiplied by 6 since 2010, indicating a new trend of theses procedures. Outpatient stays presents several advantages for the patient and for the health system: decrease of the psychological stress, higher satisfaction, minimization of the personal and domestic activity interruption, less exposure to nosocomial infections, decrease of global costs, increase of the population rate which can be treated. However, very few data report the experience of outpatient orthognathic surgery in France and the factors associated with its success or failure.

The choice of ambulatory versus complete hospitalization is decided during preoperative consultation by the surgeon in agreement with the patient. The classic surgical and anesthetic protocol of orthognathic surgery is applied whatever the type of hospitalization. The data are collected from the patient medical record (electronic patient record, orthognathic follow-up form, anesthetic sheet) and from a patient quality of life questionnaire. There is no modification of the usual follow-up, patients are seen at D-8 which is the end-study visit.

ELIGIBILITY:
Inclusion Criteria:

* all patients treated by an orthognathic surgery in Toulouse Teaching Hospital, having given an oral agreement

Exclusion Criteria:

* patient refusal
* inability to understand the information relative to the procedure, the care and the surgical suites
* American Society of Anesthesiology (ASA) Score>=3
* Severe eating disorders
* Pregnant woman

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Are not excluded from the study the minor patients, for reasons of collection bias: the population benefiting from an orthognathic surgery is carried out mainly on an adolescent population at the end of growth, to exclude these patients would therefore be a major bias to conducting the study and analyzing the results.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Rate of outpatient-to-inpatient shifts after an orthognathic procedure | 1 day
  An outpatient procedure is considered to have been converted into a traditional hospitalization if there is no discharge the same evening (D0) and therefore the patient has been transferred to a traditional hospitalization unit.
  The procedure is considered to have been performed on an outpatient basis if there was an outpatient discharge the same evening (J0)

SECONDARY OUTCOMES:
Outpatient rate | 1 day
  Rate of orthognathic procedures realized in ambulatory among all the scheduled procedures
Causes justifying the shift for patients expected outpatients | 1 day
  Causes like : pain, nausea-vomiting, slumber, anxiety, logistics)
Factors associated with a conversion in inpatient hospitalization among the patients planned in ambulatory | 1 day
  Demographic characteristics: age, sex or like Estimated amount of bleeding
Factors associated with the duration of hospitalization among the hospitalized patients on an inpatient basis | 1 day
  Total duration of intervention (intubation - extubation)
Score of the first 24 hours surgical outcome questionnaire | 1 day
  The questionnaire rating each adverse effect from 0 (no discomfort) to 4 (very important discomfort)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lauwers, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No